CLINICAL TRIAL: NCT01745432
Title: Assessment of the Manageability and Safety of ADBLOCK Adhesion Barrier System in Laparoscopic Gynaecological Surgery
Acronym: ADBEE
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Terumo Europe N.V. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: T201E4
Record Dates: First submitted 2012-08-16; First posted 2012-12-10 (Estimated); Last update posted 2016-07-06 (Estimated); Status verified 2016-07

CONDITIONS: UTERINE MYOMAS
Keywords: ADBLOCK; Adhesion Barrier System; laparoscopic surgery; myomectomy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ADBLOCK +laparoscopic surgery (Experimental): Adhesion Barrier System is site-specific sprayable adhesion barrier gel administered on the surgical field to reduce risk of adhesion formation.
  Interventions: Device: ADBLOCK
- laparoscopic surgery (No Intervention): Laparoscopic surgery only without use of adhesion barrier

INTERVENTIONS:
Device: ADBLOCK — Laparoscopic surgery
  Other Names: Adhesion Barrier System
  Arms: ADBLOCK +laparoscopic surgery

SUMMARY:
Adhesions are the most frequent complication of abdominopelvic surgery. They are internal scar tissues which form as a result of surgery which may abnormally join together what were once separate tissues and organs.

This study will assess the safety and usability of anti-adhesion agent (gel) when used after laparoscopic surgery.

The study will enroll 30 patients, (randomised 2:1) with safety primary endpoint (adverse events in ADBLOCK and surgery only group) assessed at 28 days

DETAILED DESCRIPTION:
Title: Assessment of the Manageability and Safety of ADBLOCK Adhesion Barrier System in Laparoscopic Gynaecological surgery

Design: Randomised controlled study to assess the safety, manageability and usability of ADBLOCK when used as an adjunct to laparoscopic surgery for the primary removal of ('virgin') myomas in women wishing to improve pregnancy outcomes.

Use of ADBLOCK will be assessed against laparoscopic surgery alone in 30 patients (randomised 2:1 ADBLOCK/surgery) with a pneumoperitoneum ≤90minutes.

Clinical Site Locations:

* Oldenburg, Germany
* Neuss, Germany
* Berlin, Germany

Patient Population: Women who have not completed their family planning and who are undergoing primary ('virgin') laparoscopic myomectomy with an aim to improve pregnancy outcomes.

ELIGIBILITY:
Inclusion Criteria:

* Female
* 18-45 years
* Indication for laparoscopic myomectomy according to the medical standard
* Negative pregnancy test before study entry
* Using adequate forms of contraception for 12 weeks following surgery (e.g. oral contraceptive pill, condom, no sexual intercourse)
* In good health including an ASA (American Society of Anesthesiologists) score of 2 or less
* No clinically significant and relevant abnormalities as evaluated by satisfactory medical assessment
* Planned de novo removal of myoma (includes mural and combination of mural and pedunculated myoma)
* Willing, able and likely to fully comply with study procedures and restrictions
* Given written, personally signed and dated informed consent to participate in the study as approved by the Institutional Review Board/Ethics Committee of the respective Clinical Study Site.

Exclusion Criteria:

* Pre-Operative Exclusion Criteria:
* Women who have completed their family planning
* Current pregnancy including ectopic pregnancy
* Breastfeeding
* 6 weeks post-partum
* Participation in another clinical study currently or within the last 30 days prior to enrolment
* SGOT, SGPT and/or bilirubin > 20% above the upper range of normal and considered clinically significant
* BUN and creatinine > 30% above the upper range of normal and considered clinically significant
* Concurrent use of systemic corticosteroids, antineoplastic agents and/or radiation
* Previous radiation therapy
* Diabetes
* Clinically relevant haemochromatosis, hepatic, renal, autoimmune, lymphatic, haematological or coagulation disorders
* Active pelvic or abdominal infection, or other infection with fever (>38°C)
* Extensive keloid scarring
* Known allergy to starch-based polymers
* Known or suspected intolerance or hypersensitivity to the study materials (or closely related compounds) or any of the stated ingredients -Additional surgical procedure non-obstetrics and gynaecology (non- OB/GYN) planned to be performed during the laparoscopic procedure

  ->4 myoma larger than 2 cms on preoperative ultrasound screen
* Largest myoma < 2 cms or > 8 cms diameter on pre-operative screen -GNRH agonist/antagonist treatment (except oral contraceptive - combined oestrogen/progesterone) in the 4 weeks prior to study
* Prior surgery for myoma
* Previous bowl surgery, excluding appendectomy
* Prior intra-abdominopelvic adhesive complications Intraoperative Exclusion Criteria
* Clinical evidence of cancer
* Clinical evidence of pregnancy including ectopic pregnancy
* Clinical evidence of rectovaginal endometriosis
* Clinical evidence of endometriosis American Fertility Society (AFS) class III or IV
* Use, during this procedure, of any approved or unapproved product or strategy for the purpose of preventing adhesion formation including use of O2 enhanced insufflation
* If the procedure needs to be performed by a laparotomy (decision made after laparoscopy has commenced) the patient must be withdrawn
* Any unplanned surgery which involves opening of the bowel or urinary tract
* Where hysteroscopy is required and it cannot be delayed until after removal of fibroid
* Only pedunculated fibroids
* Extensive pelvic adhesions (AFS severe adhesion score) or frozen pelvis
* Adhesions that would require lysing during planned myomectomy surgery Other than inconsequential filmy adhesions that do not require specific lysing to access operative site
* If pneumoperitoneum exceeds 90 minutes duration the patient will be assessed as a separate surgical covariate group for secondary endpoints only
* Use of fibrin glue
* Detection of myoma which are not suitable for surgery during the study procedure

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2012-08; Primary Completion 2015-08 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Safety as evaluated by assessment of adverse events in ADBLOCK and surgery only group | up to 28 days
  The rate of adverse events will be compared in treatment arm and control arm

SECONDARY OUTCOMES:
Postoperative recovery | up to 28 days
Safety as evaluated by assessment of adverse events in ADBLOCK and surgery only group | up to 24 months
Pain | before discharge, 7d, 14d, 1mo, 3mo, 6mo, 12mo, 24mo
Unanticipated device-related adverse events | before discharge, 7d, 14d, 1mo, 3mo, 6mo, 12mo, 24mo
Pregnancy (in women seeking to become pregnant) | 3mo, 6mo, 12mo, 24mo
Menstrual Cycle | 1m, 3mo, 6mo, 12mo, 24mo
Miscarriage | 1mo, 3mo, 6mo, 12mo, 24mo
Procedure related hospital readmission | 7d,14d, 1mo, 3mo, 6mo, 12mo, 24mo
Impact of covariates / Including length of pneumoperitoneum | before discharge, 7d,14d, 1mo, 3mo, 6mo, 12mo, 24mo

CONTACTS AND LOCATIONS:
Overall Officials: Rudy-Leon De Wilde, MD PhD, Principal Investigator — Pius Krankenhaus Oldenburg
Locations (3):
- Germany (3):
  - Klinik für Minimal Invasive Chirurgie, Berlin
  - Johanna Etienne Krankenhaus Neuss, Neuss
  - Pius Krankenhaus Oldenburg, Oldenburg